CLINICAL TRIAL: NCT01679327
Title: Study of Bevacizumab Plus Chemotherapy in Patients With Metastatic Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, yihebali chi, associated professor, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WY0524
Record Dates: First submitted 2012-08-18; First posted 2012-09-06 (Estimated); Last update posted 2012-09-06 (Estimated); Status verified 2012-09

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Oxaliplatin; Capecitabine; Leucovorin; Fluorouracil; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bevacizumab plus chemotherapy（XELOX or FOLFOX） (Experimental): Bevacizumab plus XELOX (Bevacizumab 7.5mg/kg d1;Xeloda 2g/m2 d1-14 divided into two times;Oxaliplatin 130mg/m2 d1;repeated in 21 days) Bevacizumab plus FOLFOX (Oxaliplatin 85mg/ m2 ivgtt d1;CF 200mg/ m2 ivgtt d1;Bevacizumab 5mg/kg ivgtt d1 5-FU 400mg /m2 ivgtt d1;5-FU 2400mg/m2 CIV 48h;repeated in 14 days)
  Interventions: Drug: Oxaliplatin; Drug: Xeloda; Drug: Calcium folinate (CF); Drug: 5-FU; Drug: Bevacizumab

INTERVENTIONS:
Drug: Oxaliplatin
  Other Names: Eloxatin
Drug: Xeloda
  Other Names: Capetabine
Drug: Calcium folinate (CF)
  Other Names: Calcium folinate
Drug: 5-FU
Drug: Bevacizumab
  Other Names: Avastin

SUMMARY:
This study evaluates the relationship of biomarker expression and efficacy of bevacizumab plus chemotherapy in patients with unresectable/metastatic colorectal cancer. Before the treatment, the investigators detect the VEGF-A,VEGF-C,VEGF-D,VEGFR-1,VEGFR-2,VEGFR-3 expression in tumor tissue by IHC and detect those protein expression level in plasma by ELISA. After at least 6 weeks treatment, the investigators detect again VEGF-A,VEGF-C,VEGF-D expression level in plasma by ELISA. The aim of the study is to identify whether those biomarkers could predict Bevacizumab efficacy.

ELIGIBILITY:
Inclusion Criteria:

* More than 18-years old,male or female
* Pathologically approved as unresectable/metastatic colorectal cancer
* KPS > 70% or ECOG 0-2
* HGB > 80 g/L, NEUT ≥ 1.5x109 /L, PLT ≥ 80x109 /L; CR < 1.5 x Upper normality，
* TB < 1.5 X Upper normality，AST or ALT < 2.5 x Upper normality.
* Signed consent

Exclusion Criteria:

* Other malignancies simultaneously except in situ cervix or nonmelanoma skin cancer
* Pregnancy or in lactation
* HGB < 80 g/L, NEUT < 1.5x109 /L, PLT < 80x109 /L; CR ≥ 1.5 x Upper normality， TB ≥ 2.5 X Upper normality，AST or ALT ≥2.5 x Upper normality，AKP ≥ 2.5 X Upper normality

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-03; Primary Completion 2014-06 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | 36 months
  During the chemotherapy,all the patients demonstrate CT scan or MR to evaluate tumor response to therapy every two cycles.According to RECIST 1.1,tumor response was recorded.

SECONDARY OUTCOMES:
progression free survival | 36 months
  The start time point was defined as when patients receive the first cycle chemotherapy.The end time point was defined as When tumor response to therapy was evaluated as PD according to RECIST 1.1 or patients die for any reason.
overall survival | 36 months
  From the time patients receive the first cycle chemotherapy to the time they die for any reason.
Number of Participants with Adverse Events | 36 months
  Every cycle we demonstrate routine blood test,routine urine test,routine stool test,blood biochemical test.We recommend patients take blood pressure at least twice a week during the therapy.If needed,patients also need have electrocardiogram test and echocardiography.We will evaluate the toxicity according to CTCAE4.0

CONTACTS AND LOCATIONS:
Overall Officials: Yihebali Chi, Doctor, Principal Investigator — Chinese Academy of Medical Sciences; Jinwan WANG, Study Director — Chinese Academy of Medical Sciences
Locations (1):
- Cancer Institute&Hospital Chinese Academy of Medical Sciences, Beijing, China